CLINICAL TRIAL: NCT01997632
Title: Phase 1 Study on the Safety and Reactogenicity of a Single Dose of Monovalent High-dose Inactivated Poliovirus Type 2 Vaccine (m-IPV2 HD) Given Intramuscularly Compared to Standard Trivalent Inactivated Poliovirus Vaccine (IPV) in Healthy Adults
Acronym: IPV-004
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2013/914; 2013-004598-29 (EudraCT Number)
Record Dates: First submitted 2013-11-22; First posted 2013-11-28 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Poliomyelitis
Keywords: Poliomyelitis; Vaccine
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- control vaccine: Imovax Polio® (Active Comparator)
  Interventions: Biological: a single dose of monovalent high-dose inactivated poliovirus type 2 vaccine (m-IPV2 HD)
- investigational vaccine (Experimental)
  Interventions: Biological: a single dose of the standard trivalent inactivated poliovirus vaccine (IPV)(Imovax Polio®).

INTERVENTIONS:
Biological: a single dose of monovalent high-dose inactivated poliovirus type 2 vaccine (m-IPV2 HD) — a single dose m-IPV2 HD (study vaccine), 0,5ml
  Arms: control vaccine: Imovax Polio®
Biological: a single dose of the standard trivalent inactivated poliovirus vaccine (IPV)(Imovax Polio®). — a single 0.5 ml dose Imovax Polio (control vaccine)
  Arms: investigational vaccine

SUMMARY:
The purpose of this study is to investigate if the study vaccine, m-IPV2 HD (vaccine that only contains polio serotype 2 in high dose), is as safe as the standard IPV Imovax (that contains the 3 serotypes of polio). This safety evaluation will be done in young adults.

If the study vaccine appears to be safe, it will be tested at a later stage in the target group (infants and children) to evaluate the immunogenicity of the vaccine. After all, the purpose is to use the study vaccine in the future to protect young children against Polio serotype 2. Disease with Polio type 2 indeed recently re-appeared, so vaccination of young children to come to a complete eradication of Polio is needed. The standard use of Imovax to protect against Polio serotype 2 would be too expensive. Therefore, a monovalent Polio vaccine containing only serotype 2 (= the vaccine that will be evaluated in this study), has been developed.

The duration of the study will be approximately 6 months. 120 subjects between 18 and 45 years of age will participate in Belgium.

During the study there will be 2 groups of subjects. Subjects will be assigned by chance to one of these groups. One group will receive one single injection of the study vaccine m-IPV2 HD (which contains only serotype 2), the other group will receive one single injection of the standard polio vaccine IPV, Imovax (which contains the 3 serotypes).

After this vaccination, there will be a follow-up period of 6 months. Subjects will be asked to come to the study centre one more time for the second visit (on Day 8, which is 7 days after the first visit). They will also receive 2 follow-up phone calls for approximately one month and 6 months after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-45 years of age
* Subjects born in Belgium or any other country where mandatory polio vaccination is performed.
* Written informed consent obtained from the subject.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  1. has practiced adequate contraception for 30 days prior to vaccination, and
  2. has a negative pregnancy test on the day of vaccination, and
  3. has agreed to continue adequate contraception for 2 months after vaccination.

Exclusion Criteria:

* Participation in another clinical trial.
* Any polio vaccine within 6 months before study inclusion.
* Any other vaccination in the period starting 14 days before administration of study vaccine and ending 28 days after administration of the study vaccine.
* Previous severe reaction after vaccination with polio vaccine.
* Known hypersensitivity to one or more components of the vaccine.
* Uncontrolled, clinically significant neuro-psychiatric, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic or endocrine disease.
* Subjects with an history of malignant disease (cancer)
* Known human immunodeficiency virus (HIV) positivity or other immune deficiency or immune suppressive treatment or auto-immune disease. For corticosteroids, a prednisone dose of <20 mg/day, or equivalent, is allowed. Inhaled and topical corticosteroids are allowed.
* Acute disease and/or fever (higher or equal to 37.5°C, measured orally) at the time of enrolment. Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory tract infection) without fever may be enrolled at the discretion of the investigator.
* Pregnant or lactating female. Subject who, in the opinion of the investigator, is unlikely to comply with the protocol or is inappropriate for any other reason.
* Known hypersensitivity to one or more components of the vaccine.
* Uncontrolled, clinically significant neuro-psychiatric, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic or endocrine disease.
* Subjects with an history of malignant disease (cancer)
* Known human immunodeficiency virus (HIV) positivity or other immune deficiency or immune suppressive treatment or auto-immune disease. For corticosteroids, a prednisone dose of <20 mg/day, or equivalent, is allowed. Inhaled and topical corticosteroids are allowed.
* Acute disease and/or fever (higher or equal to 37.5°C, measured orally) at the time of enrolment. Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory tract infection) without fever may be enrolled at the discretion of the investigator.
* Pregnant or lactating female.
* Subject who, in the opinion of the investigator, is unlikely to comply with the protocol or is inappropriate for any other reason.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
the safety of a single dose of m-IPV2 HD and licensed trivalent IPV | 4 weeks
  To assess the safety of a single dose of m-IPV2 HD and licensed trivalent IPV in healthy adults based on the incidence of serious and severe adverse events (AEs) within 4 weeks of vaccine administration.
the reactogenicity of a single dose of m-IPV2 HD and licensed trivalent IPV | 7 days
  To assess the reactogenicity of a single dose of m-IPV2 HD and licensed trivalent IPV in healthy adults based on the incidence of solicited local and general AEs within 7 days of vaccine administration.

SECONDARY OUTCOMES:
the safety of a single dose of m-IPV2 HD and licensed trivalent IPV | 6 months
  To assess the safety of a single dose of m-IPV2 HD and licensed trivalent IPV in healthy adults based on the incidence of serious AEs within 6 months of vaccine administration.

CONTACTS AND LOCATIONS:
Overall Officials: Geert Leroux-Roels, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Oost-Vlaanderen, Belgium